CLINICAL TRIAL: NCT04958148
Title: High Sodium Intake, Gut Microbiome and Blood Pressure Control
Brief Title: Salt and Gut Study
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1612471
Record Dates: First submitted 2021-05-21; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled trial. Half the participants will be in placebo arm, the other half will be in salt arm.
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High sodium (Experimental): Subjects will be counseled to consume a diet with 2,300 mg/d sodium which they will supplement with pills containing salt to achieve an intake of 4,300 mg/d sodium for 4 weeks.
  Interventions: Dietary Supplement: Salt pills
- Placebo (Placebo Comparator): Subjects will be counseled to consume a diet with 2,300 mg/d sodium and will supplement with taking placebo pills for 4 weeks.
  Interventions: Dietary Supplement: Placebo pills

INTERVENTIONS:
Dietary Supplement: Salt pills — Subjects will supplement salt pills with meals.
  Arms: High sodium
Dietary Supplement: Placebo pills — Subjects will supplement placebo pills with meals.
  Arms: Placebo

SUMMARY:
High sodium intake is a significant risk factor for hypertension. Recently, animal studies connect high sodium intake to the gut-immune axis and highlight the gut microbiome as a potential therapeutic target to counteract salt-sensitive conditions and hypertension. The objective of this project is to determine the effects of high salt intake on gut microbiota composition and gut intestine barrier integrity, leading to increased BP in humans. The investigators also hypothesize that high salt intake affects the gut microbiome in a sex-specific manner. In this pilot study, The investigators also test whether telehealth or in-person nutritional coaching help to decrease dietary sodium intake and improve diet quality

DETAILED DESCRIPTION:
The investigators will conduct a randomized, double-blind, placebo-controlled trial in normotensive and stage 1 hypertensive drug naïve participants (age 18-50 years, equal distribution of blacks and whites, and males and females, BP <140/90 mmHg). The average intake of sodium in the American diet is 3,400 mg per day. The average recommended dose is 2,300 mg per day. Eligible participants will be enrolled and provided with one-hour in-person/telehealth nutritional counseling at the GPI to reduce their sodium intake by 1,100 mg per day to achieve the sodium intake of 2,300 mg/day. Participants will then be randomized to receive either placebo or salt pills of 2,000 mg per day for four weeks while continuously receiving weekly telehealth nutritional counseling. The salt group's sodium intake will be 4,300 mg per day, while the sodium intake in the placebo group will be 2,300 mg per day. Participants will have a follow-up visit at six months after the 4-week sodium intervention. Participants will be tested four times (Figure 1). Participants will receive the first 1-hour in-person/telehealth nutrition counseling at GPI (baseline) and three weekly telehealth nutrition counseling during the 4-week intervention period.

ELIGIBILITY:
Inclusion criteria:

* Aged between 18-50 years
* African Americans (AAs) or European Americans (EAs)
* BP <140/90 mmHg
* Not on any prescription medications
* Normal kidney function (eGFR ≥ 90 ml/min/1.73 m2)

Exclusion criteria:

* Pregnant or nursing
* Previous diagnosis of major cardiovascular diseases including myocardial infarction, congestive heart failure or stroke, diabetes, autoimmune, chronic liver and kidney disease
* Previous diagnosis of Crohn's disease or any other intestinal conditions
* Previous diagnosis of major lung diseases such as chronic obstructive pulmonary disease (COPD)
* Previous diagnosis of cancer
* Alcohol and drug abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota diversity using 16s rRNA Sequencing | 4 weeks
  Subjects will be provided instructions and kits on how to collect feces and saliva samples. Saliva samples will be collected on the testing day. Feces sample will be collected on the testing day if possible; if not, it will be brought back the following day. DNA will be extracted from collected feces and saliva samples using the MoBioPowerSoil kit. The V3-V5 region of the 16S rRNA will be amplified and sequenced using the Illumina MiSeq platform. The outcome variables for microbiome data will be alpha diversity, beta diversity, and overall composition.

SECONDARY OUTCOMES:
Gut intestine barrier integrity measured by non-invasive biomarkers | 4 weeks
  Gut intestine barrier function will be determined by non-invasive biomarkers. Plasma LPS, I-FABP, DAO, zonulin, IL-6, TLR4 will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgia Prevention Institute/ Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
If we can share data without risking the identity of our participants, we will plan to share.